CLINICAL TRIAL: NCT06717451
Title: PS230005 Control-IQ 1.5 Post-Approval Study
Status: Active, not recruiting | Type: Observational
Sponsor: Tandem Diabetes Care, Inc. (Industry)
Collaborators: University of California, San Diego (Other)
Responsible Party: Sponsor
Other Study IDs: TP-0017060
Record Dates: First submitted 2024-12-02; First posted 2024-12-05 (Actual); Last update posted 2025-11-12 (Actual); Status verified 2025-11

CONDITIONS: Type 1 Diabetes
Keywords: type 1 diabetes; Control-IQ; Control-IQ 1.5; Tandem; mobi; t:slim X2; automated insulin delivery
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Pediatric Postmarket Surveillance: Yes | US Export: No

GROUPS / COHORTS (1):
- Control-IQ Technology v1.5: Real-world use of Control-IQ technology v1.5 for 12 months.
  Interventions: Device: Control-IQ Technology v1.5

INTERVENTIONS:
Device: Control-IQ Technology v1.5 — Tandem t:slim X2 insulin pump or Tandem Mobi insulin pump with Control-IQ technology v1.5.
  Every month participants will receive a survey to complete assessments including any severe hypoglycemia or diabetic ketoacidosis events experienced since the prior assessment. Participants will also complete surveys related to patient reported outcomes at baseline, 6 months, and 12 months.

SUMMARY:
This 522 post-market surveillance study is a single-arm, decentralized prospective observational cohort study designed to collect safety data on Control-IQ technology v1.5 in children with type 1 diabetes ages 2 to <6 years old. Participants will use Control-IQ technology v1.5 for 12 months in the real-world setting.

DETAILED DESCRIPTION:
The study will recruit participants age 2 to <6 years old who begin Control-IQ technology v1.5 use in the real-world setting, with a goal of a minimum of 120 completers at 12 months. All enrolled participants will be monitored from baseline through 12 months following the initiation of therapy with the Control-IQ 1.5 system. The primary endpoint is the risk of diabetic ketoacidosis (DKA) and severe hypoglycemia (SH) events. Secondary outcomes include CGM time in range measurements, and patient reported outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Self-reported type 1 diabetes who have been prescribed the Control-IQ 1.5 system in the t:slim X2 or Mobi insulin pump
* Age 2 to <6 years at time of screening
* Using an insulin approved for use in the pump
* Using an iCGM sensor approved for use with the pump
* Agreement to use Control-IQ technology 1.5, and to continue use for at least 12 consecutive months after study enrollment.
* Agree to provide HbA1c result, obtained within the 6-month period prior to enrollment.
* Ability for parent/guardian to respond to alerts and alarms, and to provide basic diabetes self-management.
* Reside full-time in the United States.
* Willingness to download the t:connect Mobile application to their smartphone and keep it active throughout the study if using a Tandem t:slim X2 pump. Participants who are unable to use the t:connect mobile application must be willing to manually upload their insulin pump data to Tandem Source every three months and at the completion of the study.
* Participant's parent/guardian has read, understood and agreed to participate in the study, and has electronically signed the Informed Consent Form (ICF).

Exclusion Criteria:

* Use of any glucose-lowering therapy other than insulin.
* A medical or other condition, or medications being taken that in the investigator's judgement would be a safety concern for participation in the study.

Ages: 2 Years to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Enrollment in the study will be available to all individuals age 2 to <6 years of age at time of screening who start therapy with Control-IQ Technology v1.5.
Sampling Method: Non-Probability Sample
Enrollment: 144 (Actual)
Dates: Start 2025-01-30 (Actual); Primary Completion 2026-08-11 (Estimated); Study Completion 2026-08-11 (Estimated)

PRIMARY OUTCOMES:
Incidence Rates of Severe Hypoglycemia (SH) | 12 months
  Overall incidence rate of SH events per 100 patient years during 12 months of Control-IQ use
Incidence Rates of Diabetic Ketoacidosis (DKA) | 12 months
  Overall incidence rate of DKA events per 100 patient years during 12 months of Control-IQ use

SECONDARY OUTCOMES:
Percent Time in Range 70 - 180 mg/dL | 12 months
  CGM measured percent time in range 70 - 180 mg/dL during 12 months of Control-IQ use
Percent Time Greater Than 180 mg/dL | 12 months
  CGM measured percent time >180 mg/dL during 12 months of Control-IQ use
Percent Time Greater Than 250 mg/dL | 12 months
  CGM measured percent time >250 mg/dL during 12 months of Control-IQ use
Percent Time Less Than 70 mg/dL | 12 months
  CGM measured percent time <70 mg/dL during 12 months of Control-IQ use
Percent Time Less Than 54 mg/dL | 12 months
  CGM measured percent time <54 mg/dL during 12 months of Control-IQ use
Mean Glucose mg/dL | 12 months
  CGM measured mean glucose during 12 months of Control-IQ use

OTHER OUTCOMES:
Diabetes Impact and Satisfaction Scale (DIDS), Satisfaction Score | 12 months
  DIDS satisfaction score at baseline, and after 6 and 12 months of Control-IQ use. Score range from 0-10 with higher scores indicating better outcome.
Diabetes Impact and Satisfaction Scale (DIDS), Impact Score | 12 months
  DIDS impact score at baseline, and after 6 and 12 months of Control-IQ use. Score range from 0 -10 with lower scores indicating better outcome.
EQ-5D (inclusive of the Visual Analogue Scale (VAS)) | 12 months
  Questionnaire score at baseline, and after 6 and 12 months of Control-IQ use.
Hypoglycemia Fear Survey - Parent for Young Children Version (HFS-P-YC) | 12 months
  Questionnaire score at baseline, and after 6 and 12 months of Control-IQ use.

CONTACTS AND LOCATIONS:
Overall Officials: Jordan Pinsker, MD, Principal Investigator — Chief Medical Officer, Tandem Diabetes Care
Locations (1):
- Tandem Diabetes Care, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No